CLINICAL TRIAL: NCT01847248
Title: HSPA12B as a Potential Biomarker for Sepsis and Severe Sepsis
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, Dr., Changhai Hospital
Other Study IDs: HSPA12B-sepsis-biomarker
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Sepsis
Keywords: sepsis; biomarker; HSPA12B
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- sepsis: Patients with sepsis but not severe sepsis
- Severe sepsis: Patients with severe sepsis
- SIRS: Patients with SIRS after major orthopedics surgery
- Control: Healthy volunteers

SUMMARY:
* Molecules indicating endothelial injury may serve as biomarkers for severe sepsis because of the critical role of endothelial injury in organ dysfunction during severe sepsis.
* HSPA12B is primarily located in endothelial cells and detectable during sepsis.
* The investigators speculated that HSPA12B from endothelial cells might be correlated with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients meet the diagnostic criteria according to the grouping

Exclusion Criteria:

* patients without informed consent
* patients who were undergoing continuous renal replacement therapy before sampling
* patients with special infection induced by virus, tubercle bacillus, mycoplasma, Chlamydia, and so on

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Continuous patients with sepsis, severe sepsis, SIRS after major orthopedics surgery and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  mortality within 28 days after recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-ming Zhu, M.D., Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Changhai Hospital
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Changhai Hospital, Shanghai, China